CLINICAL TRIAL: NCT01352572
Title: Effects of Antidepressant on Postsynaptic Signal Transduction in Serotonergic System of Depressed Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Doh Kwan Kim, M.D., pHD, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002-09-08
Record Dates: First submitted 2011-04-21; First posted 2011-05-12 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Depression
Keywords: Antidepressant Response; Signal Transduction; Lymphocyte; Biomarkers; Depressed Patients; Antidepressant Drug Adverse Reaction
MeSH Terms: conditions — Depression | interventions — Paroxetine; Milnacipran; Nortriptyline; Mirtazapine; Fluoxetine; Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antidepressant response (Experimental): antidepressant response are refered the patients having a 50 ≤ Decrease rate(%) of HAM-D score
  Interventions: Drug: antidepressant response
- antidepressant non-response (Active Comparator): antidepressant non-response are refered the patients having a 50 > Decrease rate(%) of HAM-D score
  Interventions: Drug: antidepressant non-response

INTERVENTIONS:
Drug: antidepressant response — Antidepressants administration for 6 weeks under therapeutic dose responders
  Other Names: fluoxetine_Prozac; paroxetine_Paxil, Seroxat; sertraline_Zoloft; milnacipran; venlafaxine_Effexor; nortriptyline_Aventyl, Pamelor, Noritren; mirtazapine_Avanza, Zispin, Remeron
  Arms: antidepressant response
Drug: antidepressant non-response — Antidepressants administration for 6 weeks under therapeutic dose nonresponders
  Other Names: fluoxetine, paroxetine, sertraline; milnacipran, venlafaxine, nortriptyline, mirtazapine
  Arms: antidepressant non-response

SUMMARY:
The purpose of this study is to determine whether alteration of signal transduction components after antidepressant targeting, predict antidepressant responsiveness in advance before the appearance of the drug effects until 4~6 weeks after drug administration, or represent the clinical status of depressed patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether antidepressants effect on signal transduction in peripheral lymphocyte and to determine whether the signaling differences between drug responders and nonresponders predict the antidepressant response or represent the clinical status of depressed patients.

ELIGIBILITY:
Inclusion Criteria:

1. met the Diagnostic and Statistical Manual of the American Psychiatric Association (DSM-IV) criteria for MDD from the Department of Psychiatry, Sungkyunkwan University, Seoul, South Korea.
2. were 18 years of age or older, the existence of a unipolar major depressive episode as verified by DSM-III/IV criteria, at least 2 years after first episode onset, and agreement to informed consents

Exclusion Criteria:

* pregnancy
* significant medical conditions
* abnormal laboratory baseline values
* unstable psychiatric features (e.g, suicidal attempt)
* history of alcohol or drug dependence, seizure, neurological illness, or concomitant Axis I psychiatric disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2002-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Antidepressant Response at 6 weeks | 6 weeks
  Rsponse is defined as decrease rate of HAM-D score for 6week of treament is = or >50%
  Measurement Unit = responders, nonresponders

SECONDARY OUTCOMES:
Biological value at 0 and 6 weeks | 6 weeks
  Biologial value is defined as protein expression value of signaling components in peripheral lymphocyte.
  Measurement value : Optical Density(O.D), microgram/liter(ug/l)

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Kangnam, Seoul, South Korea